CLINICAL TRIAL: NCT03154996
Title: Chronic Convection Enhanced Delivery of Topotecan for Recurrent High Grade Gliomas
Brief Title: Chronic Convection Enhanced Delivery of Topotecan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey N. Bruce (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey N. Bruce, Edgar M. Housepian Professor of Neurological Surgery Research at, Dept of Neurological Surgery, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ9520; 5R01CA161404-02 (NIH)
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Gliomas
Keywords: Gliomas; Recurrent; Chronic Convection; High Grade Gliomas
MeSH Terms: conditions — Glioma; Recurrence | interventions — Topotecan; 9 alpha,11 alpha,15 alpha-trihydroxy-16-phenoxy-17,18,19,20-tetranorprosta-4,5,13-trienoic acid; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Long term CED of Topotecan (Experimental): An additional 5 patients will be treated with TPT by CED maintained for 32 days. TPT infusions will be carried out for 32 days using Synchromed II infusion pumps with the same infusion parameters and experimental conditions used in the short term studies.
  Interventions: Drug: Topotecan; Drug: Gadolinium; Device: Synchromed II infusion pumps

INTERVENTIONS:
Drug: Topotecan — Topotecan is a chemotherapeutic agent that is a topoisomerase inhibitor. TPT is administered through an externalized catheter and external microinfusion pump.
  Dose: 146 micrometers (uM)
  Other Names: Hycamtin; TPT
Drug: Gadolinium — Gadolinium is a widely available MRI contrast agent that is used routinely in clinical practice via IV administration, especially for imaging of intracranial tumors.
  Other Names: Gado
Device: Synchromed II infusion pumps — Implanted subcutaneously to facilitate chronic infusion.

SUMMARY:
The primary goal of this study is to establish, for the first time, safety of prolonged intracerebral convection enhanced delivery of chemotherapy in patients with recurrent high grade glioma (HGG). Secondary objectives will include determination of topotecan (TPT) distribution and radiographic tumor response with prolonged continuous intracerebral convection-enhanced delivery (CED).

DETAILED DESCRIPTION:
Malignant gliomas are among the most pernicious of human tumors - locally invasive and universally recurrent, with recurrence usually occurring within two centimeters of the original resection cavity. Although numerous chemotherapeutic drugs demonstrate significant anti-tumor activity in preclinical studies, the efficacy in clinical trials has been dismal because systemic delivery fails to achieve therapeutic drug levels in tumor cells due to various factors including limited blood-brain barrier permeability and systemic toxicity.

Convection-enhanced delivery (CED) is a method of regional drug delivery that circumvents this problem. Phase 1 clinical trial has shown that a potent topoisomerase inhibitor, topotecan (TPT), can be safely and effectively delivered by CED into patients with recurrent malignant gliomas. This study will expand on these clinical results to address two current limitations to the clinical application of CED: 1) A reliable method for non-invasively monitoring drug distribution throughout the tumor and brain does not exist; and 2) Duration of CED therapy has been limited to short-term infusions secondary to the use of externalized infusion pumps.

The hypothesis is that extended chronic local-regional delivery of TPT is safe, effective and feasible in patients with recurrent gliomas. TPT will be directly and chronically delivered into the tumor and surrounding brain by CED through subcutaneously implanted pumps while innovating a methodology for monitoring the drug distribution through non-invasive imaging. This strategy will overcome the limitations of chemotherapy as currently used in the treatment of gliomas, and may be applicable to other central nervous system (CNS) diseases currently limited by drug delivery barriers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a recurrent malignant glioma (World Health Organization (WHO) grade III-IV), including recurrent glioblastoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma, and anaplastic ependymoma. Stereotactic biopsies will be performed to confirm this diagnosis prior to initiating the treatment.
* Patients with tumors of the brain must have been previously treated with surgical resection, external beam radiation, and temozolomide chemotherapy.
* An magnetic resonance (MR) scan must be obtained within 30 days of enrollment and must demonstrate an enhancing mass without significant mass effect. Tumors must be less than 32 cc in total volume. The lesion must be stereotactically accessible.
* Patients must have demonstrated evidence of increasing contrast enhancement on MR or computed tomography (CT) imaging while on stable or increasing dose of steroid.
* Karnofsky performance score of greater than or equal to 60.
* Men and women of childbearing potential must practice birth control. Women of child bearing potential must have a urine pregnancy test within 7 days of study entry.
* Patients must possess the ability to give Informed Consent.
* Patients must be willing to and medically capable of undergoing the surgical operation.
* There is no upper age limit. Patients at extreme upper end of the age spectrum will not be automatically excluded, but will be carefully scrutinized to determine their suitability for this procedure.
* Patients must be at least 18 years old.
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes: ≥3,000/ cells per microliter of blood (mcL)
  * Absolute neutrophil count: ≥1,500/mcL
  * Platelets: ≥100,000/mcL
  * Total bilirubin: within normal institutional limits
  * aspartate aminotransferase (AST) (SGOT)/alanine aminotransferase (ALT) (SGPT): ≤2.5 × institutional upper limit of normal
  * Creatinine: within normal institutional limits OR
  * Creatinine clearance: ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

Exclusion Criteria:

* Patients with diffuse subependymal or cerebral spinal fluid (CSF) disease.
* Patients with tumors involving the cerebellum or both cerebral hemispheres.
* Patients with an active infection requiring treatment or having an unexplained febrile illness.
* Patients who are known HIV, Hepatitis B or Hepatitis C positive. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with topotecan. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with systemic diseases which may be associated with unacceptable anesthetic/operative risk.
* Patients who have previously received systemic topotecan for their tumor
* Patients who are not able to receive an MRI scan.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to topotecan, other topoisomerase inhibitors or gadolinium compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Dose at which all patients have had no greater than grade 2 adverse reactions | Up to 29 days
  This is designed to measure the safety of prolonged intracerebral convection enhanced delivery of chemotherapy in patients.

SECONDARY OUTCOMES:
Clinical toxicity rate | Up to 29 days
  This is defined by the number of serious adverse events occuring, which is projected to be ≤ 5% at 23-29 days. A clinical toxicity rate that exceeds 20% will be considered unacceptable for this procedure.
Change in radiographic tumor response | Baseline, 6 weeks post-treatment
  Tumor response to TPT will be investigated by MRI scan.
Progression free survival (PFS) | Every 3-6 months, up to 5 years
  The length of time during and after the treatment of disease that a patient lives with the disease but it does not get worse. Patients will be contacted every 3-6 months, up to 5 years, by phone until death.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bruce, MD, Principal Investigator — jnb2@cumc.columbia.edu
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Spinazzi EF, Argenziano MG, Upadhyayula PS, Banu MA, Neira JA, Higgins DMO, Wu PB, Pereira B, Mahajan A, Humala N, Al-Dalahmah O, Zhao W, Save AV, Gill BJA, Boyett DM, Marie T, Furnari JL, Sudhakar TD, Stopka SA, Regan MS, Catania V, Good L, Zacharoulis S, Behl M, Petridis P, Jambawalikar S, Mintz A, Lignelli A, Agar NYR, Sims PA, Welch MR, Lassman AB, Iwamoto FM, D'Amico RS, Grinband J, Canoll P, Bruce JN. Chronic convection-enhanced delivery of topotecan for patients with recurrent glioblastoma: a first-in-patient, single-centre, single-arm, phase 1b trial. Lancet Oncol. 2022 Nov;23(11):1409-1418. doi: 10.1016/S1470-2045(22)00599-X. Epub 2022 Oct 13. PMID 36243020
- See also: Herbert Irving Comprehensive Cancer Center clinical trials online search tool — http://hiccc.columbia.edu/clinicaltrials/